CLINICAL TRIAL: NCT07171164
Title: Motivate Vaccinate Activate: An Effectiveness-Implementation Trial to Assess the Impact of a Multi-Component Community-Based Intervention to Increase RSV Vaccine Uptake Among Latino Older Adults
Brief Title: A Study to Evaluate Community-Based Measures to Increase RSV Vaccine Use Among Latino Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Mission Language Vocational School (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Motivate Vaccinate Activate; R01MD019749 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Older Adults Without Any Specific Clinical Condition; Social Networks; RSV Immunization; Vaccine Uptake
Keywords: RSV; RSV vaccine; Social networks; Counseling; Healthy adults
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Motivate Aim: CHW text message reminders and counseling (Experimental)
  Interventions: Behavioral: Motivate Aim: CHW text message reminders and counseling
- Motivate Aim: CHW text message reminders only (Active Comparator)
  Interventions: Behavioral: Motivate Aim: CHW text message reminders only
- Activate Aim: CHW text message reminders and counseling (Experimental)
  Interventions: Behavioral: Activate Aim: CHW text message reminders and counseling
- Activate Aim: CHW text message reminders only (Active Comparator)
  Interventions: Behavioral: Activate Aim: CHW text message reminders only

INTERVENTIONS:
Behavioral: Motivate Aim: CHW text message reminders and counseling — Participants receive both text message reminders and a counseling session, along with information about RSV and the vaccine, to encourage RSV vaccine uptake.
  Arms: Motivate Aim: CHW text message reminders and counseling
Behavioral: Motivate Aim: CHW text message reminders only — Participants receive text message reminders along with information about RSV and the RSV vaccine to encourage vaccine uptake, but do not receive the counseling intervention
  Arms: Motivate Aim: CHW text message reminders only
Behavioral: Activate Aim: CHW text message reminders and counseling — Participants receive both text message reminders and a counseling session, along with information about RSV and the vaccine, to encourage discussion of RSV vaccine uptake among older adults in their social networks
  Arms: Activate Aim: CHW text message reminders and counseling
Behavioral: Activate Aim: CHW text message reminders only — Participants receive text message reminders along with information about RSV and the vaccine to encourage discussion of RSV vaccine uptake among older adults in their social networks, but do not receive the counseling intervention
  Arms: Activate Aim: CHW text message reminders only

SUMMARY:
In collaboration with community-based organizations, this study will focus on increasing RSV vaccine use among Latinos. The study will determine how effective community health worker counseling and text-message approaches are to (1) increase RSV vaccine use among older adults (Motivate phase) and (2) encourage younger adults to discuss RSV vaccination with their older friends and family members (Activate phase).

DETAILED DESCRIPTION:
In this type 1 hybrid-implementation study, the investigators will utilize a well-established community-academic partnership to achieve multiple aims. In the Motivate phase, the study will randomize 400 Latino older adults to community health worker (CHW) counseling and text message nudges vs. CHW delivered RSV vaccine vs. text-message nudges alone. The primary outcome in the Motivate phase is RSV vaccine uptake. In the Activate phase, using a parallel design, investigators will randomize 350 Latino adults (18-49 years) to CHW 'activation' counseling to encourage them to discuss RSV vaccine with people over 50 and older in their network plus text-message nudges, vs. text-message nudges alone. The primary outcome for the Activate phase is the average proportion of older adults in participants' social network with whom they discussed RSV vaccination. Interventions in both phases will be adapted using community-based participatory research principles.

ELIGIBILITY:
Motivate Aim Inclusion Criteria:

* Age 50 years or older
* Self-identify as Latino/a/x and/or indigenous groups from Latin America
* Eligible for RSV vaccination per current CDC/ACIP recommendations
* Fluent in Spanish or English
* Has not received the RSV vaccine
* Has a cell phone
* Lives or works in San Francisco or Daly City
* Able to provide informed consent

Motivate Aim Exclusion Criteria:

* Intent to move outside of San Francisco or Daly City in the next year
* Nursing home resident
* Household member participating in Aim 1 or 2
* Unable to provide consent

Motivate Aim Inclusion Criteria:

* Age 18-49 years
* Self-identify as Latino/a/x and/or indigenous groups from Latin America
* Fluent in English or Spanish
* Has >1 family member or friend 50 years or older who they have seen or spoken to for >15 minutes in the last 6 months and who lives in the United States

Activate Trial Exclusion Criteria:

* Household member enrolled in Aim 1 or 2
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Motivate Aim Primary Outcome - RSV Vaccine Uptake | 60 days from study enrollment
  RSV vaccine uptake at 60 days per California Immunization Registry (CAIR) or per medical record
Activate Aim Primary Outcome - Proportion of Contacts with whom RSV Vaccination Discussed | 60 days after study enrollment
  Self-reported average proportion of social network contacts 50 years or older with whom participant discussed RSV vaccination at 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Carina Marquez, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackerson B, Tseng HF, Sy LS, Solano Z, Slezak J, Luo Y, Fischetti CA, Shinde V. Severe Morbidity and Mortality Associated With Respiratory Syncytial Virus Versus Influenza Infection in Hospitalized Older Adults. Clin Infect Dis. 2019 Jul 2;69(2):197-203. doi: 10.1093/cid/ciy991. PMID 30452608
- [Background] Juhn YJ, Wi CI, Takahashi PY, Ryu E, King KS, Hickman JA, Yao JD, Binnicker MJ, Natoli TL, Evans TK, Sampathkumar P, Patten C, Luyts D, Pircon JY, Damaso S, Pignolo RJ. Incidence of Respiratory Syncytial Virus Infection in Older Adults Before and During the COVID-19 Pandemic. JAMA Netw Open. 2023 Jan 3;6(1):e2250634. doi: 10.1001/jamanetworkopen.2022.50634. PMID 36662530
- [Background] Zheng Z, Warren JL, Shapiro ED, Pitzer VE, Weinberger DM. Estimated incidence of respiratory hospitalizations attributable to RSV infections across age and socioeconomic groups. Pneumonia (Nathan). 2022 Oct 25;14(1):6. doi: 10.1186/s41479-022-00098-x. PMID 36280891
- [Background] Mahmud SM, Xu L, Hall LL, Puckrein G, Thommes E, Loiacono MM, Chit A. Effect of race and ethnicity on influenza vaccine uptake among older US Medicare beneficiaries: a record-linkage cohort study. Lancet Healthy Longev. 2021 Mar;2(3):e143-e153. doi: 10.1016/S2666-7568(20)30074-X. Epub 2021 Feb 18. PMID 36098112
- [Background] McLaughlin JM, Khan F, Begier E, Swerdlow DL, Jodar L, Falsey AR. Rates of Medically Attended RSV Among US Adults: A Systematic Review and Meta-analysis. Open Forum Infect Dis. 2022 Jun 17;9(7):ofac300. doi: 10.1093/ofid/ofac300. eCollection 2022 Jul. PMID 35873302

DOCUMENTS (3):
  • Study Protocol (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT07171164/Prot_000.pdf
  • Informed Consent Form: Aim 2 Motivate Informed Consent Form (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT07171164/ICF_001.pdf
  • Informed Consent Form: Aim 3 Activate Informed Consent Form (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT07171164/ICF_002.pdf